CLINICAL TRIAL: NCT02867397
Title: A Phase 1, Open-Label, Non-Randomized, Dose-Finding, Safety and Tolerability Study of Orally Administered Teysuno (S-1) in Combination With Epirubicin and Oxaliplatin in Patients With Advanced Solid Tumors
Brief Title: Study of Teysuno (S-1) Combined With Epirubicin and Oxaliplatin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Disphar International B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1119
Record Dates: First submitted 2016-08-11; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Patients With Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — tegafur-gimeracil-oteracil; S 1 (combination); Epirubicin; Oxaliplatin

ARMS (1):
- Teysuno (S1) in combination with epirubicin and oxaliplatin (Other)
  Interventions: Drug: Teysuno (S1) in combination with epirubicin and oxaliplatin

INTERVENTIONS:
Drug: Teysuno (S1) in combination with epirubicin and oxaliplatin

SUMMARY:
The goal of the current study was to investigate the safety and determine the maximum tolerated dose (MTD) of S-1 in combination with oxaliplatin and epirubicin in patients with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Had given written informed consent.
2. Was ≥18 years of age.
3. Had advanced or metastatic solid tumor(s) for which no established curative therapy exists.
4. Had received any number of prior therapies for advanced or metastatic disease.
5. Was able to take medications orally.
6. Had ECOG performance status 0 or 1 on Cycle 1, Day 1
7. Had a life expectancy of at least 3 months.
8. Had LVEF ≥ the LLN for the institution.
9. Had serum troponin T and CPK-MB values ≤ ULN for the institution.
10. Had adequate organ function as defined by the following criteria:

    1. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5 x ULN; if liver function abnormalities were due to underlying liver metastasis, AST (SGOT) and ALT (SGPT) ≤5 x ULN.
    2. Total serum bilirubin of ≤1.5 x ULN.
    3. Absolute neutrophil count of ≥1,500/mm3 (ie, ≥1.5 x 109/L by International Units [IU]) (excluding measurements obtained within 7 days after administration of granulocyte colony-stimulating factor (G-CSF).
    4. Platelet count ≥100,000/mm3 (IU: ≥100 x 109/L) (excluding measurements obtained within 7 days after transfusion).
    5. Hemoglobin value of ≥9.0 g/dL (excluding measurements obtained within 7 days after transfusion).
    6. Creatinine clearance ≥60 mL/min based on calculated creatinine clearance or 24-hour urine collection.
11. Was willing and able to comply with scheduled visits, treatment plan, lab tests and other study procedures.

Exclusion Criteria:

1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

   1. Major surgery within prior 4 weeks (the surgical incision should be fully healed prior to study drug administration).
   2. Radiotherapy within prior 4 weeks.
   3. >25% of marrow-bearing bone radiated (Pre-Amendment 3).
   4. Any chemotherapy within prior 3 weeks.
   5. Previously received oxaliplatin or S-1.
   6. Previously received epirubicin with cumulative dose >350 mg/m2 (patients who have received epirubicin with cumulative dose ≤350 mg/m2 as adjuvant therapy are allowed to enroll).
   7. Extensive prior exposure to other anthracycline or anthracenedione agents (ie, prior cumulative doxorubicin exposure of ≥450 mg/m2 or prior mitoxantrone exposure of >100 mg/m2)
   8. Received trastuzumab (cardiotoxic agent) within prior 24 weeks.
   9. Any investigational agent received either concurrently or within the last 30 days.
   10. Current enrollment in another interventional clinical study.
2. Has a serious illness or medical condition(s) including, but not limited to, the following:

   1. Known brain metastasis or leptomeningeal metastasis.
   2. Known acute systemic infection.
   3. Myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack, pulmonary embolism, or deep vein thrombosis within the last 12 months.
   4. Symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV (see Appendix E).
   5. Ongoing cardiac dysrhythmias (≥Grade 2), atrial fibrillation (any grade), or prolongation of QTc interval (>450 msec for males; >470 msec for females).
   6. Hypertensive crisis or severe hypertension that is not controlled.
   7. Chronic nausea, vomiting, or diarrhea considered to be clinically significant in the opinion of the Investigator.
   8. ≥Grade 1 peripheral neuropathy.
   9. Recent hemoptysis, coagulopathy and other bleeding disorders considered by the Investigator to be clinically significant.
   10. Known nephrotic syndrome (proteinuria >2 g/24 hours).
   11. Known clinically significant interstitial lung disease or pulmonary fibrosis.
   12. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
   13. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.
3. Is receiving concomitant treatment with the following drugs that may interact with S-1:

   1. Sorivudine, brivudine, uracil, eniluracil, cimetidine, folinate/folinic acid, and dipyridamole (may enhance S-1 activity).
   2. Nitroimidazoles, including metronidazole and misonidazole (may enhance S-1 activity)
   3. Methotrexate (may enhance S-1 activity)
   4. Clozapine (may increase risk and severity of hematologic toxicity with S-1)
   5. Allopurinol (may diminish S-1 activity).
   6. Phenytoin (S-1 may enhance phenytoin activity).
   7. Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 activity).
4. Is receiving concomitant treatment with the following drugs that may interaction with epirubicin:

   1. Cimetidine (may increase the area under the plasma concentration-time curve [AUC] of epirubicin).
   2. Dexverapamil (may alter the pharmacokinetics of epirubicin).
   3. Quinine (may accelerate the initial distribute on of epirubicin from blood into the tissues and may have an influence on the red blood cells partitioning of epirubicin).
   4. Interferon alfa-2b (may cause a reduction in both the terminal elimination half-life and the total clearance of epirubicin).
5. Is a pregnant or lactating female.
6. Has known hypersensitivity to 5-FU, epirubicin, oxaliplatin or other platinum compounds.
7. Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients). Contraceptive measures must be taken by both male and female patients during and up to 6 months after stopping treatment with S-1.

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The highest dose level at which less than 33% of the patients experienced a dose-limiting toxicity (DLT) during Cycle 1. | 21 days